CLINICAL TRIAL: NCT06304415
Title: Investigating The Prevalence and Clinical Significance of Elevated Lipoprotein(a) Blood Levels in Hospital Staff
Brief Title: Elevated Lipoprotein(a) in Hospital Staff
Acronym: LPACO
Status: Recruiting | Type: Observational
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Loh Wann Jia, Primary Investigator and Consultant Endocrinologist., Changi General Hospital
Other Study IDs: CIRB2023/2651
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-08

CONDITIONS: Hypercholesterolemia; Lipoprotein Types--Lp System Lp(A) Hyperlipoproteinemia; Cardiovascular Diseases
MeSH Terms: conditions — Hypercholesterolemia; Lipoprotein Types--Lp System Lp(A) Hyperlipoproteinemia; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood are collected to measure lipoprotein(a) concentrations, genetic variants and biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Working General Population: Consenting hospital staff are recruited to this study. Blood test and questionnaires are taken at baseline. Prospective follow-up of cardiovascular events are undertaken.

SUMMARY:
The objective of this study is to investigate the prevalence of elevated Lp(a) in the working general population.

DETAILED DESCRIPTION:
The objective of this study is to investigate the prevalence of elevated lipoprotein(a) concentrations and distribution of lipoprotein(a) in a working general population. This is a prospective study investigating the association of lipoprotein(a) with cardiovascular markers and outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Any healthcare workers working in healthcare settings (regardless of PHI and/or private setting) aged 21 and above OR family member such as father, mother, siblings, grandparents, spouse and children aged 12 and above of recruited staff with high Lpa ≥120nmol/l
2. Study team members can also be recruited because we are trying to find the prevalence of elevated Lp(a)

Exclusion Criteria:

1. Inability to provide informed consent.
2. Pregnant women.
3. Prisoner

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Working general population
Sampling Method: Non-Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2035-12-01 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Distribution and prevalence of elevated Lipoprotein(a) | 3 years
  Investigate the distribution lipoprotein(a) and prevalence of elevated lipoprotein(a) concentrations in various ethnicities.

SECONDARY OUTCOMES:
Correlation of lipoprotein(a) with cardiovascular outcomes | 10 years
  Observational study to assess the correlation of degree of elevation of lipoprotein(a) with cardiovascular outcomes prospectively.
Genetic variants of lipoprotein(a) and cardiovascular outcomes atherosclerotic events | 10 years
  Assess the association of genetic variants of lipoprotein(a) with the measured lipoprotein(a) concentrations in various ethnicities, and prospectively assess the association of these genetic variants with cardiovascular outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Loh Wann Jia, Principal Investigator — Singhealth Foundation
Locations (1):
- Clinical Trials & Research Unit, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loh WJ, Watts GF. Detection strategies for elevated lipoprotein(a): will implementation let the genie out of the bottle? Curr Opin Endocrinol Diabetes Obes. 2023 Apr 1;30(2):94-102. doi: 10.1097/MED.0000000000000789. Epub 2022 Dec 5. PMID 36468313
- [Background] Loh WJ, Chang X, Aw TC, Phua SK, Low AF, Chan MY, Watts GF, Heng CK. Lipoprotein(a) as predictor of coronary artery disease and myocardial infarction in a multi-ethnic Asian population. Atherosclerosis. 2022 May;349:160-165. doi: 10.1016/j.atherosclerosis.2021.11.018. Epub 2021 Nov 26. PMID 34887076
- [Background] Loh WJ, Chan DC, Mata P, Watts GF. Familial Hypercholesterolemia and Elevated Lipoprotein(a): Cascade Testing and Other Implications for Contextual Models of Care. Front Genet. 2022 Apr 27;13:905941. doi: 10.3389/fgene.2022.905941. eCollection 2022. PMID 35571022
- [Background] Nestel P, Loh WJ, Ward NC, Watts GF. New Horizons: Revival of Lipoprotein (a) as a Risk Factor for Cardiovascular Disease. J Clin Endocrinol Metab. 2022 Nov 23;107(11):e4281-e4294. doi: 10.1210/clinem/dgac541. PMID 36108076
- [Background] Kronenberg F, Mora S, Stroes ESG, Ference BA, Arsenault BJ, Berglund L, Dweck MR, Koschinsky M, Lambert G, Mach F, McNeal CJ, Moriarty PM, Natarajan P, Nordestgaard BG, Parhofer KG, Virani SS, von Eckardstein A, Watts GF, Stock JK, Ray KK, Tokgozoglu LS, Catapano AL. Lipoprotein(a) in atherosclerotic cardiovascular disease and aortic stenosis: a European Atherosclerosis Society consensus statement. Eur Heart J. 2022 Oct 14;43(39):3925-3946. doi: 10.1093/eurheartj/ehac361. PMID 36036785